CLINICAL TRIAL: NCT05418088
Title: Phase I Clinical Trial of Anti-CD19/20/22 Chimeric Antigen Receptor T Cells for Treatment of Relapsed or Refractory Lymphoid Malignancies (Non-Hodgkin Lymphoma, Acute Lymphoblastic Leukemia, Chronic Lymphocytic Leukemia, B-Prolymphocytic Leukemia)
Brief Title: Genetically Engineered Cells (Anti-CD19/CD20/CD22 CAR T-cells) for the Treatment of Relapsed or Refractory Lymphoid Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sumithira Vasu (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Sumithira Vasu, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSU-21170; NCI-2022-02972 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); R01CA276374 (NIH)
Record Dates: First submitted 2022-05-16; First posted 2022-06-14 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Recurrent Acute Lymphoblastic Leukemia; Recurrent B Acute Lymphoblastic Leukemia; Recurrent B-Cell Prolymphocytic Leukemia; Recurrent Chronic Lymphocytic Leukemia; Recurrent High Grade B-Cell Lymphoma; Recurrent Indolent Non-Hodgkin Lymphoma; Recurrent Non-Hodgkin Lymphoma; Recurrent Transformed Chronic Lymphocytic Leukemia; Refractory Acute Lymphoblastic Leukemia; Refractory B Acute Lymphoblastic Leukemia; Refractory B-Cell Prolymphocytic Leukemia; Refractory Chronic Lymphocytic Leukemia; Refractory High Grade B-Cell Lymphoma; Refractory Indolent Non-Hodgkin Lymphoma; Refractory Non-Hodgkin Lymphoma; Refractory Transformed Chronic Lymphocytic Leukemia; Refactory Childhood Acute Lymphoblastic Leukemia; Refractory Childhood Non-Hodgkin Lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Leukemia, Prolymphocytic, B-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin | interventions — Cyclophosphamide; fludarabine phosphate; Biopsy; Blood Component Removal; Leukapheresis; Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort A (lymphodepletion; anti-CD19/CD20/CD22 CAR-T cells) (Experimental): LYMPHODEPLETIVE REGIMEN: Patients receive cyclophosphamide IV over 60 minutes on day -6 and fludarabine IV over 30 minutes on days -5 to -3 in the absence of disease progression or unacceptable toxicity.
  CAR T-CELL THERAPY: Patients receive anti-CD19/CD20/CD22 CAR-T cells IV over 5-30 minutes on day 0.
  Patients undergo ECHO or MUGA and may undergo tissue biopsy during screening, undergo apheresis on study, and undergo bone marrow biopsy and aspiration and blood sample collection throughout the study.
  Interventions: Biological: Anti-CD19/CD20/CD22 CAR T-Cells; Drug: Cyclophosphamide; Drug: Fludarabine Phosphate; Procedure: Echocardiography; Procedure: Multigated Acquisition Scan; Procedure: Biopsy; Procedure: Pheresis; Procedure: Bone Marrow Aspiration and Biopsy; Procedure: Biospecimen Collection
- Cohort B (lymphodepletion, anti-CD19/CD20/CD22 CAR-T cells) (Experimental): LYMPHODEPLETIVE REGIMEN: Patients receive cyclophosphamide IV over 60 minutes on day -6 and fludarabine IV over 30 minutes on days -5 to -3 in the absence of disease progression or unacceptable toxicity.
  CAR T-CELL THERAPY: Patients receive anti-CD19/CD20/CD22 CAR-T cells IV over 5-30 minutes on day 0 and 7.
  Patients undergo ECHO or MUGA and may undergo tissue biopsy during screening, undergo apheresis on study, and undergo bone marrow biopsy and aspiration and blood sample collection throughout the study.
  Interventions: Biological: Anti-CD19/CD20/CD22 CAR T-Cells; Drug: Cyclophosphamide; Drug: Fludarabine Phosphate; Procedure: Echocardiography; Procedure: Multigated Acquisition Scan; Procedure: Biopsy; Procedure: Pheresis; Procedure: Bone Marrow Aspiration and Biopsy; Procedure: Biospecimen Collection
- Cohort C (lymphodepletion, anti-CD19/CD20/CD22 CAR-T cells) (Experimental): LYMPHODEPLETIVE REGIMEN: Patients receive cyclophosphamide IV on days -6 and -5 and fludarabine IV on days -6 to -3 in the absence of disease progression or unacceptable toxicity.
  CAR T-CELL THERAPY: Patients receive anti-CD19/CD20/CD22 CAR-T cells IV over 5-30 minutes on day 0 and 7.
  Patients undergo ECHO or MUGA and may undergo tissue biopsy during screening, undergo apheresis on study, and undergo bone marrow biopsy and aspiration and blood sample collection throughout the study.
  Interventions: Biological: Anti-CD19/CD20/CD22 CAR T-Cells; Drug: Cyclophosphamide; Drug: Fludarabine Phosphate; Procedure: Echocardiography; Procedure: Multigated Acquisition Scan; Procedure: Biopsy; Procedure: Pheresis; Procedure: Bone Marrow Aspiration and Biopsy; Procedure: Biospecimen Collection

INTERVENTIONS:
Biological: Anti-CD19/CD20/CD22 CAR T-Cells — Given IV
  Other Names: Anti-CD19/20/22 Chimeric Antigen Receptor T-Cells; CD19/CD20/CD22-targeted CAR-T Cells
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Procedure: Echocardiography — Undergo echocardiography
  Other Names: EC
Procedure: Multigated Acquisition Scan — Undergo MUGA scan
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Procedure: Biopsy — Undergo tissue biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Pheresis — Undergo apheresis
  Other Names: Apheresed; apheresis; Blood Component Removal; Collection; Apheresis/Leukapheresis; Hemapheresis
Procedure: Bone Marrow Aspiration and Biopsy — Undergo bone marrow aspiration and biopsy
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection

SUMMARY:
This phase I trial tests the safety, side effects and best infusion dose of genetically engineered cells called anti-CD19/CD20/CD22 chimeric antigen receptor (CAR) T-cells following a short course of chemotherapy with cyclophosphamide and fludarabine in treating patients with lymphoid cancers (malignancies) that have come back (recurrent) or do not respond to treatment (refractory). Lymphoid malignancies eligible for this trial are: non-Hodgkin lymphoma (NHL), acute lymphoblastic leukemia (ALL), chronic lymphocytic leukemia (CLL), and B-prolymphocytic leukemia (B-PLL). T-cells (a type of white blood cell) form part of the body's immune system. CAR-T is a type of cell therapy that is used with gene-based therapies. CAR T-cells are made by taking a patient's own T-cells and genetically modifying them with a virus so that they are recognized by a group of proteins called CD19/CD20/CD22 which are found on the surface of cancer cells. Anti-CD19/CD20/CD22 CAR T-cells can recognize CD19/CD20/CD22, bind to the cancer cells and kill them. Giving combination chemotherapy helps prepare the body before CAR T-cell therapy. Giving CAR-T after cyclophosphamide and fludarabine may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the safety of the treatment of relapsed/refractory non-Hodgkin lymphoma, relapsed/refractory chronic lymphocytic leukemia, refractory B-prolymphocytic leukemia and relapsed/refractory acute lymphoblastic leukemia with chimeric antigen receptor T cells targeting CD19/20/22 and to find the recommended phase II dose for this cellular therapy.

SECONDARY OBJECTIVES:

I. To describe the safety profile of the infusion of CAR-T cells targeting CD19/20/22 in relapsed/refractory Non-Hodgkin lymphoma, relapsed/refractory chronic lymphocytic leukemia, refractory B-prolymphocytic leukemia and in relapsed/refractory acute lymphoblastic leukemia.

II. To describe the toxicities related to infusion of CAR-T cells targeting CD19/20/22.

III. To describe the overall response rate and complete response rate of relapsed B cell malignancies treated with CAR-T cells targeting CD19/20/22.

IV. To describe the overall and progression free survival of patients with relapsed lymphoma, CLL, B-PLL and ALL treated with anti-CD19/20/22 CAR-T cells.

EXPLORATORY OBJECTIVES:

I. To describe the persistence of anti-CD19/20/22 CAR-T cells, measured by flow cytometry and quantitative polymerase chain reaction (qPCR).

II. To describe the T cell subpopulations of the anti-CD19/20/22 CAR-T cell product before infusion.

III. To describe the changes in anti-CD19/20/22 CAR-T cells after infusion and their correlation with disease response and adverse events.

IV. To investigate the correlation between changes in cytokine plasma concentrations and changes in anti-CD19/20/22 CAR-T cell subpopulations over time.

V. To investigate proteomic changes in anti-CD19/20/22 CAR-T cell subpopulations over time.

VI.To investigate whether antigen escape occurs in patients treated with anti-CD19/20/22 CAR-T.

OUTLINE: This is a phase I dose-escalation study of anti-CD19/CD20/CD22 CAR-T cells. Patients with NHL with lesions =< 5 cm, indolent lymphomas, CLL (without Richter's transformation), or B-PLL are assigned to Cohort A. Patients with ALL, CLL (with Richter's transformation), NHL with lesions > 5 cm and/or lymphoblastic lymphoma, or NHL with circulating lymphoma cells are assigned to Cohort B.

COHORT A:

LYMPHODEPLETIVE REGIMEN: Patients receive cyclophosphamide intravenously (IV) over 60 minutes on day -6 and fludarabine IV over 30 minutes on days -5 to -3 in the absence of disease progression or unacceptable toxicity.

CAR T-CELL THERAPY: Patients receive anti-CD19/CD20/CD22 CAR-T cells IV over 5-30 minutes on day 0.

Patients undergo echocardiography (ECHO) or multigated acquisition scan (MUGA) and may undergo tissue biopsy during screening, undergo apheresis on study, and undergo bone marrow biopsy and aspiration and blood sample collection throughout the study.

COHOHRT B:

LYMPHODEPLETIVE REGIMEN: Patients receive cyclophosphamide IV over 60 minutes on day -6 and fludarabine IV over 30 minutes on days -5 to -3 in the absence of disease progression or unacceptable toxicity.

CAR T-CELL THERAPY: Patients receive anti-CD19/CD20/CD22 CAR-T cells IV over 5-30 minutes on day 0 and 7.

Patients undergo ECHO or MUGA and may undergo tissue biopsy during screening, undergo apheresis on study, and undergo bone marrow biopsy and aspiration and blood sample collection throughout the study.

COHORT C:

LYMPHODEPLETIVE REGIMEN: Patients receive cyclophosphamide IV on days -6 and -5 and fludarabine IV on days -6 to -3 in the absence of disease progression or unacceptable toxicity.

CAR T-CELL THERAPY: Patients receive anti-CD19/CD20/CD22 CAR-T cells IV over 5-30 minutes on day 0 and 7.

Patients undergo ECHO or MUGA and may undergo tissue biopsy during screening, undergo apheresis on study, and undergo bone marrow biopsy and aspiration and blood sample collection throughout the study.

After completion of study treatment, patients in Cohort A are followed up on days 1-7, 14, 21, 30, 60, 90, at months 6, 24, 36, 48, and 60, and then annually for 6-15 years. Patients in Cohort B and Cohort C are followed up on days 9, 14, 21, 30, 60, 90, at months 6, 24, 36, 48, and 60, and then annually for 6-15 years.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects with relapsed or refractory non-Hodgkin lymphoma with lesions =< 5 cm, indolent lymphomas, chronic lymphocytic leukemia without Richter's transformation, or B-prolymphocytic leukemia (Cohort A)
* OR adult subjects with lymphoid blast crisis, acute lymphoblastic leukemia, chronic lymphocytic leukemia with Richter's transformation, non-Hodgkin lymphoma with lesions > 5 cm and/or lymphoblastic lymphoma, or non-Hodgkin lymphoma with circulating lymphoma cells, B-Prolymphocytic leukemia with lesions > 5 cm (not including splenomegaly (Cohort B).
* OR Pediatric subjects with Acute Lymphoblastic Leukemia or Non-Hodgkin Lymphoma
* Subjects must have been treated with at least two lines of therapy. Disease must have either progressed after the last regimen or presented failure to achieve complete remission with the last regimen. B-PLL is defined as having greater than 55% prolymphocytes in the peripheral blood
* Subjects with relapsed/refractory CLL after at least 2 prior lines of appropriate therapy and must have previously received an approved BTK inhibitor and venetoclax
* Subjects with refractory high-grade B-cell lymphoma who relapse within 12 months of autologous stem cell transplant
* Subjects with relapsed/refractory B-prolymphocytic leukemia who received at least 1- 2 prior lines of appropriate therapy and who have failed or are ineligible for allogeneic stem cell transplant
* Subjects with relapsed/refractory acute B-lymphoblastic leukemia who received at least 2 prior lines of appropriate therapy or who have failed or are ineligible for allogeneic stem cell transplant.
* The patient's lymphoid malignancy must be positive for at least one target antigen (CD19 and/or CD20 and/or CD22), either by immunohistochemistry or flow cytometry analysis on the last biopsy available or peripheral blood for circulating disease.
* Patients who received blinatumomab or inotuzumab are eligible.
* Patients who received prior CAR T-cells are eligible, (commercial CD 19 CAR-T cells or dual CAR-T cells), if it has been at least 30 days since previous CAR T cell therapy and <5% of circulating levels of CD3+ cells express the prior CAR by flow cytometry.
* Age >= 2 years
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2. For patients < 16 years, Performance score Lansky >= 50
* Total bilirubin =< 1.5 times the institutional upper limit of normal for age
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) =< 3 X institutional upper limit of normal for age
* Alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 X institutional upper limit of normal for age
* Creatinine clearance more than or equal to 50 ml/min calculated by the Cockcroft - Gault formula, or by Schwartz formula for patients < 18 years
* Subjects must have adequate pulmonary function as defined as pulse oximetry >= 92% on room air
* Subjects must have adequate cardiac function as defined as left ventricular ejection fraction >= 40% in the most recent echocardiogram
* Absolute lymphocyte count > 100/uL
* Subjects (or legal guardians) must have the ability to understand and the willingness to sign a written informed consent document
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use a contraceptive method with a failure rate of < 1% per year during the treatment period and for at least 6 months after the Anti-CD19/20/22 CAR-T cell infusion
* A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (< 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus). Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptive s that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices
* The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm
* With female partners of childbearing potential, men must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of < 1% per year during the treatment period and for at least 6 months after the Anti-CD19/20/22 CAR-T cell infusion. Men must refrain from donating sperm during this same period
* With pregnant female partners, men must remain abstinent or use a condom during the treatment period and for at least 6 months after the human anti-CD19 CAR-T cell infusion to avoid potential embryonal or fetal exposure. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.

Exclusion Criteria:

* Autologous transplant within 6 weeks of planned CAR-T cell infusion
* Allogeneic stem cell transplant or donor lymphocyte infusion within 2 months of planned CAR-T cell infusion and patients must be off immunosuppressive agents. Patients with live vaccines given 28 days prior to lymphodepletion (LD) chemotherapy will be excluded
* Active graft versus host disease
* Active central nervous system or meningeal involvement by lymphoma or leukemia. Subjects with untreated brain metastases/central nervous system (CNS) disease will be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. Patients with a history of CNS or meningeal involvement must be in a documented remission by CSF evaluation and contrast-enhanced magnetic resonance imaging (MRI) imaging for at least 90 days prior to registration
* Active malignancy, other than non-melanoma skin cancer or carcinoma in situ (e.g.cervix, bladder, breast). Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial (e.g.

Low Gleason score prostate Cancer)

* A minimum of 28 days must have elapsed between prior treatment with investigational agent(s) and the day of lymphocyte collection
* Human immunodeficiency virus (HIV)-seropositive patients are allowable, however must be on effective anti-retroviral therapy with undetectable viral load within 6 months of enrollment to be eligible for this trial
* Subjects with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, pulmonary abnormalities or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or breastfeeding women are excluded from this study because CAR-T cell therapy may be associated with the potential for teratogenic or abortifacient effects. Women of childbearing potential must have a negative serum pregnancy test. Because there is an unknown, but potential risk for adverse events in nursing infants secondary to treatment of the mother with CAR-T cells, breastfeeding should be discontinued. These potential risks may also apply to other agents used in this study
* Evidence of myelodysplasia or cytogenetic abnormality indicative of myelodysplasia on any bone marrow biopsy prior to initiation of therapy
* Patients with a positive hepatitis B core antibody or surface antigen are at high risk for hepatitis B virus (HBV) reaction and will require entecavir/tenofivir prophylaxis or serial hepatitis B (Hep B) PCR monitoring at the direction of an infectious disease specialist. Duration of prophylaxis to correspond with detection of Anti-CD19/20/22 CAR T cells/viral vector copies in serum or continued evidence of B-cell aplasia such as reduced intravenous immunoglobulin therapy (IVIG) levels. No antiviral prophylaxis is indicated with hepatitis C positivity with negative PCR
* Patients with history of clinically relevant CNS pathology such as epilepsy, seizure disorders, paresis, aphasia, uncontrolled cerebrovascular disease, severe brain injuries, dementia and Parkinson's disease
* History of autoimmune disease (i.e. rheumatoid arthritis, systemic lupus erythematosus) with requirement of immunosuppressive medication within 6 months
* Live vaccines given in 28 days prior to lymphodepleting chemotherapy

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2022-06-30 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Recommended phase II dose of anti-CD19/CD20/CD22 CAR-T cells for each study group (Cohort A, Cohort B, and Cohort C) | Up to 30 days after CAR T-cell infusion

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 12 months after completion of study treatment
  Will be evaluated with descriptive statistics for the frequencies of adverse events of different grades.
Overall response rate | Up to 15 years
  Will be evaluated with descriptive statistics with proportions used to describe response rates.
Complete response rate | Up to 15 years
  Will be evaluated with descriptive statistics with proportions used to describe response rates.
Overall survival | Up to 15 years
  Will be calculated using Kaplan Meier method, comparisons between groups will be done using the log rank test.
Progression-free survival | From entry onto study until lymphoma progression or death from any cause, assessed up to 15 years
  Will be calculated using Kaplan Meier method, comparisons between groups will be done using the log rank test.

OTHER OUTCOMES:
Correlation between cytokine serum concentrations and disease response | Up to 15 years
  Will be analyzed with descriptive statistics, including evaluations of median, minimum and peak values. Area under the curve (AUC) will be used as a measure of cytokine secretion. Comparisons will be done between responding and non-responding patients using the Mann - Whitney test for quantitative variables and Fisher's exact test for categorical variables. The Wilcoxon test will be used to evaluate the changes in cytokine concentrations. Correlations between quantitative variables will be done with Spearman's correlation test, whereas correlation between categorical variables will be done using Fisher's exact test.
Presence of measurable CAR-T cells | Up to 12 months
  Will be analyzed with descriptive statistics, including evaluations of median, minimum and peak values. Area under the curve (AUC) will be used as a measure of CAR-T cell expansion and persistence. Comparisons will be done between responding and non-responding patients using the Mann - Whitney test for quantitative variables and Fisher's exact test for categorical variables. The Wilcoxon test will be used to evaluate CAR-T cell expansion and changes in T cell phenotype over time. Correlations between quantitative variables will be done with Spearman's correlation test, whereas correlation between categorical variables will be done using Fisher's exact test.
Correlation between CD19/20/22 expression on disease response | Up to 15 years
  Will be analyzed with descriptive statistics, including evaluations of median, minimum and peak values. Correlations between quantitative variables will be done with Spearman's correlation test, whereas correlation between categorical variables will be done using Fisher's exact test.

CONTACTS AND LOCATIONS:
Overall Officials: Sumithira Vasu, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Nationwide Children's Hospital, Columbus, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu